CLINICAL TRIAL: NCT02551393
Title: A Cluster-randomized Study on the Risk Assessment and Management Program for Home Blood Pressure Monitoring in Population With Inadequate Health Literacy
Brief Title: Enhancing the Risk Assessment and Management Program by Promotion of Self-blood Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Sau-nga Fu, Ph D Student, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KW/EX-15-115(88-14)
Record Dates: First submitted 2015-09-09; First posted 2015-09-16 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
Keywords: Home Blood Pressure Monitoring; Health literacy; Blood Pressure control
MeSH Terms: conditions — Hypertension | interventions — Educational Status; 4-(2-(4-hydroxybenzyl)-phenoxy)-N-methylbutylamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Doctors and Nurses in intervention clinic will receive 1 hour briefing + education on the background, scientific basis and detail of the program during lunch time. People from intervention clinics will be invited to attend 2 x 2 hours education group (15-30 subjects / group) ran by clinic nurses and doctors. You will be educated on basic knowledge, management and drug for hypertension in the first session. In the 2nd session, a certified valid Home BP device will be loaned to you for 6-9 months and you will be taught to perform home Blood pressure monitoring, record and response to the BP reading accordingly. Upon completion of session 2, you will be arranged for nurse individual follow up after 4-8 weeks to see their progress and monitoring
  Interventions: Behavioral: Home Blood Presssure Monitoring, Education
- Control Group (No Intervention): Usual Care of hypertension in primary care clinic

INTERVENTIONS:
Behavioral: Home Blood Presssure Monitoring, Education — Doctors and Nurses in intervention clinic will receive 1 hour briefing + education on the background, scientific basis and detail of the program during lunch time. People from intervention clinics will be invited to attend 2 x 2 hours education group (15-30 subjects / group) ran by clinic nurses and doctors. You will be educated on basic knowledge, management and drug for hypertension in the first session. In the 2nd session, a certified valid Home BP device will be loaned to you for 6-9 months and you will be taught to perform home BP monitoring, record and response to the BP reading accordingly. Upon completion of session 2, you will be arranged for nurse individual follow up after 4-8 weeks to see their progress and monitoring
  Other Names: HBPM
  Arms: Intervention Group

SUMMARY:
Clinical Trial: The investigators aims at comparing providing validated home BP device, followed by group education of self-management of hypertension as well as self-BP monitoring and appropriate medication in response to home BP reading, followed by nurse follow up with usual care, which may possibly improve patients with uncontrolled hypertensions drug adherence, and therefore improve their BP level in primary care setting. The investigators will invite total 270 patients from 5 general outpatient clinic (GOPCs) to participate the trial.

Qualitative study: The investigators would also like to evaluate patients' view and operational concerns on self BP monitoring by individually interviewing 30 selected patients with uncontrolled hypertension

DETAILED DESCRIPTION:
Background Recent oversea randomized control trials have proven effectiveness of lowering clinic and home BP if uncontrolled hypertensive patients were taught to perform home BP monitoring properly with validated BP device. Patients were taught to response to home BP reading (e.g. follow drug regime, or doctor adjust drug according to patients' home BP record)

Study design 1. Prospective cluster randomized control trial, 2. Qualitative individual interview

Aims The investigators aims at comparing providing validated home BP device, followed by group education of self-management of hypertension as well as self-BP monitoring and appropriate medication in response to home BP reading, followed by nurse follow up with usual care, which may possibly improve older adults with uncontrolled hypertension drug adherence, and therefore improve their BP level in a primary care setting. The investigators would also like to evaluate patients' view and operational concerns on self BP monitoring

Subjects Adult Chinese on hypertensive treatment more than 12 months with uncontrolled hypertension by mean clinic BP measurement on the day of recruitment. Uncontrolled hypertension is defined as BP > 140/90mmHg in subjects age < 80; and BP > 150/90mmHg in subjects age≥80. You will be invited to participate if you are willing and capable to perform self-home BP monitoring on daily basis.

Sample size 270 (45 people from each clinic); 30 people for qualitative interview

Assignment 3 clinics will be randomly assigned to intervention clinic while the other 2 will be randomly assigned to the control clinic (usual care)

Intervention(s) Doctors and Nurses in intervention clinic will receive 1 hour briefing + education on the background, scientific basis and detail of the program during lunch time. Patients from intervention clinics will be invited to attend 2 x 2 hours education group (15-30 subjects / group) ran by clinic nurses and doctors. You will be educated on basic knowledge, management and drug for hypertension in the first session. In the 2nd session, a certified valid Home BP device will be loaned to you for 6- 9 months and you will be taught to perform home BP monitoring, record and respond to the BP reading accordingly. Upon completion of session 2, you will be arranged for nurse individual follow up after 4-8 weeks to see your progress and monitoring.

30 people with uncontrolled hypertension will be interviewed individually for their opinion on the program, management of hypertension and performance of home BP monitoring.

Outcome measures BMI (BH/ BW), Waist circumference, Clinic BP (sitting position/ standing position), Lab Test: FBS, Lipid profile, eGFR, Urine PCR, ECG Qualitative data for patient's view on home BP monitoring

Follow up duration 6-18months

ELIGIBILITY:
Inclusion Criteria:

1. Adult
2. Chinese
3. on hypertensive treatment
4. uncontrolled hypertension by mean clinic BP measurement on the day of recruitment. Uncontrolled hypertension is defined as BP > 140/90mmHg in subjects age < 80; and BP > 150/90mmHg in subjects age≥80.
5. willing and capable to perform home BP monitoring by themselves on daily basis. -

Exclusion Criteria:

1. unable to perform the home monitoring either by themselves
2. mentally incapacitated
3. arrhythmias
4. unstable angina
5. serum creatinine > 250 mmol/l
6. orthostatic hypotension
7. severe left ventricular impairment
8. severe aortic stenosis
9. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Clinic Blood Pressure control rate | 18 months
  After 18 months of treatment, to compare BP control rate in the intervention group and the control group.

SECONDARY OUTCOMES:
Proportion of subjects with normal body mass index | 18 months
  To compare the BW and BMI over time
Change of fasting blood sugar level | 18 months
  To compare the fasting blood sugar level over time
Change of low density lipoprotein level (LDL) | 18 months
  To compare the low density lipoprotein level (LDL) over time
Change in mean clinic Systolic blood pressure (SBP) intervention group when compare with control group | 6 months, 12 months and 18 months
  To comparer the SBP level over time
Change in mean clinic diastolic blood pressure DBP intervention group when compare with control group | 6 months, 12 months and 18 months
  To compare intervention group when compared with control group
Qualitative study of patients' view and experience of home blood pressure monitoring | 5 patients are interviewed before intervention, 6 weeks post-intervention, different time frame after patients' hypertension diagnosed
  Patients' experience were report in the framework of the social cognitive theory

CONTACTS AND LOCATIONS:
Overall Officials: Sau Nga FU, MBBS, Principal Investigator — Kwoloon West Cluster, Hospital Authority

REFERENCES:
- [Derived] Fu SN, Dao MC, Wong CKH, Cheung BMY. Knowledge and practice of home blood pressure monitoring 6 months after the risk and assessment management programme: does health literacy matter? Postgrad Med J. 2022 Aug;98(1162):610-616. doi: 10.1136/postgradmedj-2020-139329. Epub 2021 May 26. PMID 34039693
- [Derived] Fu SN, Dao MC, Luk W, Lam MCH, Ho ISF, Cheung SK, Wong CKH, Cheung BMY. A cluster-randomized study on the Risk Assessment and Management Program for home blood pressure monitoring in an older population with inadequate health literacy. J Clin Hypertens (Greenwich). 2020 Sep;22(9):1565-1576. doi: 10.1111/jch.13987. Epub 2020 Aug 18. PMID 32810355

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-01-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT02551393/Prot_ICF_000.pdf